CLINICAL TRIAL: NCT05018936
Title: Efficacy and Safety of Hetrombopag in Non-severe Aplastic Anemia: a Prospective Single Arm Study
Brief Title: Efficacy and Safety of Hetrombopag in Non-severe Aplastic Anemia
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Principal Investigator, Bing Han, Docter, Peking Union Medical College Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HBP-NSAA-001
Record Dates: First submitted 2021-08-19; First posted 2021-08-24 (Actual); Last update posted 2021-08-24 (Actual); Status verified 2021-08

CONDITIONS: Aplastic Anemia; Drug Effect
MeSH Terms: conditions — Anemia, Aplastic | interventions — hetrombopag

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- treatment group (Experimental): Hetrombopag would be started with 5mg/day. The dosage would be increased by 2.5mg/day every 2 weeks if the platelet count remains less than 20×10e9/L and reduced if the platelet count reaches over than 150×10e9/L. The maximum dosage is 15mg/day.
  Interventions: Drug: Hetrombopag

INTERVENTIONS:
Drug: Hetrombopag — Hetrombopag starting at 5mg/day and increased by 2.5mg/day every 2 weeks if the platelet count remains less than 20×10e9/L and reduced if the platelet count reaches over than 150×10e9/L.

SUMMARY:
This is a prospective one arm study to explore the efficacy and safety of Hetrombopag in non-severe aplastic anemia. Patients meeting the inclusion and exclusion criteria would be recruited. Treatment of Hetrombopag would be started with 5mg/day. The dosage would be increased by 2.5mg/day every 2 weeks if the platelet count remains less than 20×10e9/L and reduced if the platelet count reaches over than 150×10e9/L. The maximum dosage is 15mg/day. All patients would receive treatment for at least 6 months except that the platelet <20×10e9/L at the dosage of 15mg/day for 4 weeks or the platelet ≥200×10e9/L at the dosage of 5mg/week for 2 weeks. The hematological response rate and safety will be recorded and compared at D15, 1month, 1.5month, 2month, 3month, 4month, 5month, 6month, 8month, 10month and 1year.

ELIGIBILITY:
Inclusion Criteria:

1. Patients diagnosed to be non-severe aplastic anemia
2. Patients with platelet count < 30×109/L and have at least one of the followings: ①absolute neutrophil count < 1.5×109/L, ②platelet count < 50×109/L, ③ hemoglobin level < 100g/L
3. Patients have no response or relapsed following at least one treatment course in a period time of > 6 months of immunosuppression containing CsA or CsA+anti-thymocyte globulin (ATG);
4. Eastern Cooperative Oncology Group (ECOG) performance status 0-2;
5. Patients able to understand and comply with protocol requirements and instructions and have signed and dated informed consent.

Exclusion Criteria:

1. Congenital aplastic anemia;
2. Presence of chromosomal aberration;
3. Evidence of a clonal hematologic bone marrow disorder (MDS, AML) on cytogenetics;
4. Presence with PNH clone ≥50%;
5. Patients received HSCT before;
6. Uncontrolled infection or bleeding with standard treatment;
7. Allergic to Hetrombopag or accessories;
8. HIV, HCV or HBV active infection or liver cirrhosis or portal hypertension;
9. Patient with QTcF (Fridericia's QT correction formula) at screening <450 msec, or<480 msec with bundle branch block, as determined via the mean of a triplicate ECG and assessed at site, unstable angina pectoris, uncontrolled hypertension(>180/100mmHg)，pulmonary artery hypertension;
10. Have any concomitant malignancies within 5 years expect for local basal cell carcinoma of the skin;
11. Past history of thromboembolic event, heart attack or stroke (including anti-phospholipid antibody syndrome) and current use of anticoagulants;
12. Pregnant or nursing (lactating) woman;
13. Have attended other clinical trials within 3 months;

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2021-10-01 (Estimated); Primary Completion 2023-10-01 (Estimated); Study Completion 2023-12-01 (Estimated)

PRIMARY OUTCOMES:
ORR at 6 Months | 6 month
  Overall Response Rate (ORR) Defined as the Number of Participants Who Met the Criteria of Either Complete Response (CR) or Partial Response (PR) at 6 months

SECONDARY OUTCOMES:
ORR at 3 Months | 3 month
  ORR will be calculated after 3 months of treatment by measuring platelet, reticulocyte, neutrophil and transfusion independence.
Volume of Platelet Transfusions | 12 months
  Volume of Platelet Transfusions every month
percentage of side effects at 12 months | 12 months
  percentage of side effects would be recorded during the study and be calculated according to CTCAE 5.0 at 12 months
Percentage of patients with clonal evolution at 12 months | 12 months
  Percentage of patients with clonal evolution would be evaluated by bone marrow biopsy at 12 months follow up.

CONTACTS AND LOCATIONS:
Overall Officials: Bing Han, Master, Study Director — Peking Union Medical College Hospital
Locations (1):
- Peking Union Medical College Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: Yes
individual participant data would be accepted upon request
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: 10 years
Access Criteria: email request

REFERENCES:
- [Background] Mei H, Liu X, Li Y, Zhou H, Feng Y, Gao G, Cheng P, Huang R, Yang L, Hu J, Hou M, Yao Y, Liu L, Wang Y, Wu D, Zhang L, Zheng C, Shen X, Hu Q, Liu J, Jin J, Luo J, Zeng Y, Gao S, Zhang X, Zhou X, Shi Q, Xia R, Xie X, Jiang Z, Gao L, Bai Y, Li Y, Xiong J, Li R, Zou J, Niu T, Yang R, Hu Y. A multicenter, randomized phase III trial of hetrombopag: a novel thrombopoietin receptor agonist for the treatment of immune thrombocytopenia. J Hematol Oncol. 2021 Feb 25;14(1):37. doi: 10.1186/s13045-021-01047-9. PMID 33632264